CLINICAL TRIAL: NCT04524858
Title: A Phase 2a, Open-Label, Single-Arm Study to Investigate the Safety and Efficacy of ATI-450 for the Maintenance of Remission in Patients With Cryopyrin-Associated Periodic Syndrome (CAPS) Previously Managed With Anti-IL-1 Therapy
Brief Title: Study of ATI-450 in Patients With Cryopyrin-Associated Periodic Syndrome (CAPS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to patient enrollment challenges stemming from the COVID-19 pandemic, Aclaris has decided to focus its efforts and resources on other immuno-inflammatory diseases.
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI-450-CAPS-201
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Cryopyrin-Associated Periodic Syndrome
Keywords: Cryopyrin-Associated Periodic Syndrome; CAPS
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATI-450 (Experimental): Oral, small molecule MK2 inhibitor will be administered twice daily (BID) at a dose of 50 mg
  Interventions: Drug: ATI-450

INTERVENTIONS:
Drug: ATI-450 — Oral, small molecule MK2 inhibitor

SUMMARY:
This is a Phase 2 study to investigate the safety and efficacy of ATI-450 for the Maintenance of Remission in Patients with Cryopyrin-Associated Periodic Syndrome (CAPS) Previously Managed with Anti-IL-1 Therapy.

DETAILED DESCRIPTION:
This is a Phase 2a, Open-Label, Single-Arm Study to Investigate the Safety and Efficacy of ATI-450 for the Maintenance of Remission in Patients with Cryopyrin-Associated Periodic Syndrome (CAPS) Previously Managed with Anti-IL-1 Therapy. The study will consist of up to an 8-week screening period, a 12-week treatment period, and a 4-week safety follow-up period. The total duration of the study for patients remaining until their final follow-up assessment will be up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Familial Cold Autoinflammatory Syndrome, Muckle-Wells Syndrome, or Neonatal Onset Multisystem Inflammatory Disease. Prior agreement between the Investigator and Aclaris for study eligibility is required for patients who do not have a molecular diagnosis of NALP3 mutations available (either testing not performed, or testing performed, but negative) upon study entry. For those patients who have not been molecularly tested for NALP3 mutations, molecular testing should be performed during the study.
* Patients with a PGA score of "minimal" or less and hsCRP and SAA values within the normal range (≤10mg/L), and who are considered to have achieved that response as a result of successful anti-IL-1 therapy.
* Continuous Treatment with anti-IL1 therapy for at least 6 months.
* Able to understand and comply with study procedures and able to provide informed consent.
* Male or non-pregnant, non-nursing female patients at least 18 years of age, inclusive.

  * Female patients who are of childbearing potential must use 2 methods of highly effective contraception* - one of which must be a physical barrier- for the duration of the study and for 30 days after the last dose.
  * Male patients of childbearing potential with a female partner of childbearing potential must agree to use a condom plus another highly effective form of birth control for the duration of the study and for 90 days after the last dose.
* Female patients must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to dosing on Day 1.
* Willing and capable of taking appropriate Covid-19 risk mitigation precautions (e.g. wearing a mask in public, adhering to social distancing, etc.) as required by local, state, or federal guidelines during participation in the study.

Exclusion Criteria:

* Participation in any clinical study with an investigative agent within 12 weeks prior to entry or within 5 half-lives of the investigational agent.
* Being treated with another immuno-suppressive agent (i.e., in addition to an anti-IL-1 product) for CAPS syndrome (anti- IL-1 therapy will have been used for at least 6 months and will be stopped at study entry).
* Use of any of the following treatments within the indicated washout period prior to the baseline visit:

  * Systemic immunosuppressant or immunomodulatory therapy (e.g., etanercept, alefacept, infliximab, methotrexate) within 16 weeks prior to Visit 2 (excluding anti- IL-1 therapy for CAPS).
  * Janus Kinase (JAK) inhibitors (systemic or topical) within 4 weeks prior to Visit 2.
  * Systemic corticosteroids within 4 weeks prior to Visit 2 (Intranasal, inhaled, and topical ocular corticosteroids are allowed).
* History of being immunocompromised, including a positive HIV at screening (ELISA and Western blot) test result. [Previous treatment with anti-IL1 therapy is not an exclusion]
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody test result.
* Live vaccinations within 3 months prior to the start of the trial, or during the trial.
* History of recurrent and/or evidence of active bacterial, fungal, or viral infections.
* History or evidence of active or latent tuberculosis (TB).
* Tests performed at a central laboratory at screening that meet any of the criteria below (out of range labs may be rechecked one time, after consultation with sponsor or designee, before patient is considered a screen failure):

  * White blood cell (WBC) count <3.0×103 cells/mm3
  * Absolute neutrophil count (ANC) <1.5×103 cells/mm3
  * Lymphocyte count <0.5×103 cells/mm3
  * Platelet count <100×103 cells/mm3
  * Hemoglobin <10 g/dL
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2×upper limit of normal (ULN)
  * Total bilirubin level >2×ULN, unless patient has been diagnosed with Gilberts' disease and this is clearly documented
  * Estimated glomerular filtration rate Estimated glomerular filtration rate (eGFR), <40 mL/min/1.73m2 based on Modification of Diet and Renal Disease formula
* Any clinically significant laboratory abnormality that would affect interpretation of study data or safety of the patient's participation in the study, per the judgment of the investigator.
* Patient has clinically significant abnormal findings other than CAPS from physical examination that may affect the interpretation of study data or the safety of the patient's participation in the study, per the judgment of the investigator.
* Patient has a clinically important history of a medical disorder that would compromise patient safety or data quality, per the judgement of the investigator.
* Blood pressure (BP) levels (in supine position after at least 5 minutes rest): <90 mmHg or >140 mmHg for systolic BP or <40 mmHg or >90 mmHg for diastolic blood pressure.
* Patients with history of stroke.
* Significant cardiac disease that would affect interpretation of study data or the safety of the patient's participation in the study, per the judgment of the investigator, including recent myocardial infarction or unstable angina, or heart failure with New York Heart Association Class III or IV symptoms.
* Patients with the following screening or pre-dose ECG findings, specifically:

  * Evidence of atrial fibrillation, atrial flutter, complete right or left bundle branch block, Wolff-Parkinson-White Syndrome, or other significant rhythm disturbance
  * Evidence of acute ischemia
  * Screening or pre-dose baseline mean QTcF >450 msec for males or >470 msec for females (use of the ECG algorithm is acceptable for this purpose)
  * Personal or family history of congenital long QT syndrome or sudden death
  * Any other finding that is considered clinically significant
* A confirmed diagnosis of Covid-19 at baseline or at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gordon, Study Director — Aclaris Therapeutics
Locations (2):
- United States (2):
  - Aclaris Investigational Site, San Diego, California
  - Aclaris Investigational Site, San Francisco, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATI-450
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Due to study termination and only 1 participant being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Arm/Group | ATI-450
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to week 12
Population: as for baseline characteristics
Arm/Group | ATI-450
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 114
Description: Due to study termination and only 1 participant being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Arm/Group | ATI-450
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT04524858/Prot_SAP_001.pdf